CLINICAL TRIAL: NCT04405934
Title: A Phase III Prospective, Interventional, Cohort, Superiority Study to Evaluate the Benefit of Rapid COVID-19 Genomic Sequencing (the COVID-19 GENOMICS UK Project) on Infection Control in Preventing the Spread of the Virus in United Kingdom NHS Hospitals
Brief Title: COG-UK Project Hospital-Onset COVID-19 Infections Study
Acronym: COG-UK HOCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Public Health England (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: CTU/2020/353; 283014 (Other: IRAS); 20/EE/0118 (Other: REC reference)
Record Dates: First submitted 2020-05-07; First posted 2020-05-28 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Covid-19; Nosocomial Infection; Coronavirus; Coronavirus Infection; SARS-CoV 2
Keywords: Nosocomial Covid-19; Covid-19; Coronavirus; Infection Prevention and Control
MeSH Terms: conditions — COVID-19; Cross Infection; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Superiority model:
  1. Baseline/control phase 1 Sample collection and genomic sequencing from Covid-19 positive participants suspected of acquiring infection in hospital (suspected nosocomial Covid-19 infection where tested positive >48 hours after hospital admission) where sequencing reports not interpreted/actioned by Infection Prevention Control (IPC) site teams
  2. Site intervention phase Sample collection and genomic sequencing from Covid-19 positive participants suspected of acquiring infection in hospital where sequencing reports generated both rapid or standard and received by site IPC teams for interpretation and action
  3. Control phase 2 (prospective) Sample collection and genomic sequencing from Covid-19 positive participants suspected of acquiring infection in hospital where sequencing reports not interpreted/actioned by IPC site teams - where deemed ethical and approved by oversight committees i.e. DMEC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genomic-sequence informed IPC measures (Other): Cohort follow baseline (no report receipt), then rapid vs standard sequencing report receipt phase, then return to baseline phase (no report receipt)
  Interventions: Other: Use of virus (Covid-19) genome sequence report to inform infection prevention control procedures

INTERVENTIONS:
Other: Use of virus (Covid-19) genome sequence report to inform infection prevention control procedures — Rapid or standard (time to return to sites) receipt of virus (Covid-19) genomic sequencing reports

SUMMARY:
Hospitals are recognised to be a major risk for the spread of infections despite the availability of protective measures. Under normal circumstances, staff may acquire and transmit infections, but the health impact of within hospital infection is greatest in vulnerable patients. For the novel coronavirus that causes COVID-19, like recent outbreaks such as the SARS and Ebola virus, the risk of within hospital spread of infection presents an additional, significant health risk to healthcare workers.

Infection Prevention and Control (IPC) teams within hospitals engage in practices that minimise the number of infections acquired within hospital. This includes surveillance of infection spread, and proactively leading on training to clinical and other hospital teams.

There is now good evidence that genome sequencing of epidemic viruses such as that which causes COVID-19, together with standard IPC, more effectively reduces within hospital infection rates and may help identify the routes of transmission, than just existing IPC practice. It is proposed to evaluate the benefit of genome sequencing in this context, and whether rapid (24-48h) turnaround on the data to IPC teams has an impact on that level of benefit.

The study team will ask participating NHS hospitals to collect IPC information as per usual practice for a short time to establish data for comparison. Where patients are confirmed to have a COVID-19 infection thought to have been transmitted within hospital, their samples will be sequenced with data fed back to hospital teams during the intervention phase. A final phase without the intervention may take place for additional information on standard IPC practice when the COVID-19 outbreak is at a low level nationwide.

DETAILED DESCRIPTION:
Hospitals are recognised to be a major risk for the spread of infections despite the availability of protective measures. Under normal circumstances, staff may acquire and transmit infections, but the health impact of nosocomial infection is greatest in vulnerable patients. For COVID-19, like SARS-CoV, MERS-CoV and Ebola virus, the risk of nosocomial spread of infection presents an additional and significant health risk to healthcare workers (HCW). During epidemics, normal infection prevention and control (IPC) practice is further complicated by the difficulties of distinguishing community- and hospital-acquired infections. This can lead to erroneous identification of nosocomial transmission, involving unnecessary IPC efforts, while true nosocomial transmissions are missed thereby putting patients and HCW at increased risk.

There is now good evidence that genome sequencing of epidemic viruses, together with standard IPC, better excludes nosocomial transmissions and, depending on the virus, better identifies routes of transmission, than IPC alone1-3. To date, all studies have been retrospective. However, the development of rapid nanopore sequencing methods enables identification of potentially linked or unlinked viruses within 24-48 hours: this timescale is short enough to inform clinical IPC decisions in near-real-time. Although COVID-19 has a low mutation rate estimated at around 2.5 changes per genome per month, it is generally agreed that sufficient viral diversity now exists to identify where patient and staff infections that are apparently clustered in time and space, are in fact due to different COVID-19 genotypes4. Such information would rapidly exclude nosocomial transmission as the cause of the cluster, reduce the need for IPC intervention and provide reassurance to healthcare workers that IPC measures including personal protective equipment (PPE), had not been breached. However, confirmation of COVID-19 transmission to patients and healthcare workers may be more difficult with a single observed mutation between two genomes feasibly representing anything between one and ten transmissions. Identical genomes will not necessarily provide evidence of a link between two cases. Nonetheless by placing genotypes detected within the framework of all the genotypes detected within the hospital setting, the surrounding community and COG-UK as a whole, it may be possible to postulate nosocomial transmission where comparatively uncommon genotypes are apparently linked or cluster in time and space.

The COG-UK initiative, which aims to sequence as many COVID-19 viruses as possible across the UK thus provides an important and unique opportunity to test whether viral sequence data produced in near-real-time, in addition to providing valuable information for public health planning, could also reduce uncertainties around nosocomial transmission events, better target IPC effort, improve hospital functioning and reduce the role of hospitals as a source of infection to the community.

To address this,the investigators propose an adjunctive study, COG-UK HOCI. COG-UK HOCI will take advantage of the COG-UK design, with its mixed model of smaller sequencing hubs located close to hospitals and a large centralised hub sequencing most viruses, to identify not only whether rapid viral sequencing is useful for patient management but how time-critical this might be ; turnaround times for sequence data from the central hub are likely to be longer (5-7 days) than those from local sequencing hubs (<48 hours).

COG-UK HOCI, by defining and reporting COVID-19 genotype frequencies within its participating hospitals, as compared to those in the wider community, will also have the potential to overcome some of the inherent barriers to identifying the likely sources of HOCI. The data generated will provide as accurate as possible a picture, given the constraints of viral genetic diversity, of numbers of COVID-19 infections being acquired by nosocomial transmission and where these transmissions are occurring. While COG-UK will provide data on the utility of viral genomics for national public health planning, COG-UK HOCI will quantify the utility of the same data for local management of nosocomial infection, whether observed benefits are time dependent and deliver the best estimates of how viral sequence data can be used to quantify HOCI.

The outputs from COG-UK HOCI will further inform decisions about the likely future use of viral genome sequencing for the management of epidemics and pandemics and how it might best be organised, centralised or diversified, to deliver maximal impact.

The overarching aim of this study is to determine the utility of whole-genome sequencing to provide additional insight into hospital-onset COVID-19 infections (HOCI) which, in turn, can optimise IPC measures. In addition, the project aims to provide early data to help quantify HOCI events and where these are occurring. These will contribute to local trust level planning and to understanding of the role of HOCIs in contributing to COVID-19 outcomes and spread.

Specifically, the study will determine the role of real-time availability of COVID-19 sequence data:

* In conjunction with routine IPC data, to identify and characterise HOCI
* To identify and characterise HOCI not previously identified by routine IPC data
* To generate estimated numbers of HOCI and where these are occurring
* To identify linked HOCI and hospital outbreaks
* To identify ways to reduce the incidence of HOCI
* In optimising IPC actions, e.g. by reducing the need for extra cleaning, ward closures etc where a hospital outbreaks are excluded
* In changing workload, e.g. by reducing the need for extra cleaning, ward closures etc where a hospital outbreaks are excluded Augmenting these approaches, the investigators will measure whether the above are influenced by the time to sequence data result.

COG-UK HOCI is a phase III prospective, interventional, cohort, superiority study.

Allocation to either rapid local sequencing (c.24-48h) or lack of rapid local sequencing (i.e. via Wellcome Sanger Institute at >96h) will be dependent on the time of the study (see timelines).

Proposed study duration: 12 months; comprising 6 months of set-up, baseline data collection, interventional data collection) and up to 6 months of data cleaning, data analysis and reporting.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have confirmed COVID-19 infection and either:

  1. be a potential hospital-onset COVID-19 infection (HOCI); or
  2. potential workplace infection from COV-SARS-2 for site-based healthcare workers.
* Participants must have provided nasal swab/pharyngeal swab / combined nasal and pharyngeal swab / nasopharyngeal aspirate or broncho alveolar lavage sample for evaluation in the COG-UK project.
* Participants may be of any age to be included in study For clarity, in the above criterion a potential HOCI is an admitted patient at site with first confirmed test for COVID-19 >48 hours after admission, where they were not suspected to have COVID-19 at time of admission.

Exclusion Criteria:

- There are no exclusion criteria for COG-UK HOCI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2170 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Incidence rates of IPC-defined hospital-onset COVID-19 infection (HOCIs) | 6 months
  Incidence rate of IPC-defined HOCIs, measured as incidence rate of recorded cases per week per 100 inpatients, during each phase of the study based on case report forms.
Change in incidence rates of IPC-defined HOCIs with rapid vs standard sequencing | 6 months
  Identification of nosocomial transmission using sequencing data in potential HOCIs in whom this was not identified by pre-sequencing IPC evaluation, measured using pre- and post-sequencing case report forms for each enrolled patient during study phases in which the sequence reporting tool is in use.

SECONDARY OUTCOMES:
Incidence rates of IPC-defined hospital outbreaks | 6 months
  Incidence rate of IPC-defined hospital outbreaks, defined as cases of hospital transmission linked by location and with intervals between diagnoses of no greater than 2 weeks (relevant data extracted from case report forms), measured as incidence rate of outbreak events per week per 100 inpatients during each phase of the study.
Incidence rates of IPC+sequencing-defined hospital outbreaks | 6 months
  Incidence rate of IPC+sequencing-defined hospital outbreaks, defined by retrospective review of all available sequencing and epidemiological data for identification of transmission clusters and measured as outbreak events per week per 100 inpatients during each phase of the study.
Changes to IPC actions following viral sequence reports | 6 months
  Changes to IPC actions implemented following receipt of viral sequence report, measured using pre- and post-sequencing case report forms for each enrolled patient during study phases in which the sequence reporting tool is in use.
Recommended changes to IPC actions following viral sequence report - not implemented | 6 months
  Changes to IPC actions that would ideally have been implemented (given unlimited resources) following receipt of viral sequence report, measured using pre- and post-sequencing case report forms for each enrolled patient during study phases in which the sequence reporting tool is in use.
Health economic benefit to IPC of standard vs rapid sequencing reports | 6 months
  Health economic benefit of standard and rapid sequencing reports to IPC measured using bespoke health economic case report data comparison between baseline, standard and rapid sequencing phases.
Impact of both standard and rapid sequencing reports on number of HCW days off work | 6 months
  Number of HCW days off work measured from sampling these data points on case report forms at all study phases.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Breuer, MD, Principal Investigator — University College, London
Locations (1):
- University College London Hospitals NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The fully anonymised datasets analysed during the study will be stored on a publicly available repository. The COG-UK HOCI study to be shared on the UCL Data Repository data-sharing platform so that the data may be reused by other researchers. The protocol will also be shared.
Supporting Information: Study Protocol
Time Frame: This will be done with 6 months of public reporting of results, with data available for 5 years.
Access Criteria: Fully open access

REFERENCES:
- [Derived] Stirrup O, Blackstone J, Mapp F, MacNeil A, Panca M, Holmes A, Machin N, Shin GY, Mahungu T, Saeed K, Saluja T, Taha Y, Mahida N, Pope C, Chawla A, Cutino-Moguel MT, Tamuri A, Williams R, Darby A, Robertson DL, Flaviani F, Nastouli E, Robson S, Smith D, Loose M, Laing K, Monahan I, Kele B, Haldenby S, George R, Bashton M, Witney AA, Byott M, Coll F, Chapman M, Peacock SJ; COG-UK HOCI Investigators; COVID-19 Genomics UK (COG-UK) consortium; Hughes J, Nebbia G, Partridge DG, Parker M, Price JR, Peters C, Roy S, Snell LB, de Silva TI, Thomson E, Flowers P, Copas A, Breuer J. Effectiveness of rapid SARS-CoV-2 genome sequencing in supporting infection control for hospital-onset COVID-19 infection: Multicentre, prospective study. Elife. 2022 Sep 13;11:e78427. doi: 10.7554/eLife.78427. PMID 36098502